CLINICAL TRIAL: NCT03430921
Title: Open-label, Prospective, Multicenter Study to Evaluate the Cutera Enlighten™ Laser and a Micro-Lens Array Handpiece Attachment for the Treatment of Moderate to Severe Acne Scars
Brief Title: Evaluation of the Cutera Enlighten™ Laser With Micro-Lens Array (MLA) Handpiece Attachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-17-ML03
Record Dates: First submitted 2018-02-01; First posted 2018-02-13 (Actual); Results first posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Scarring; Acne
MeSH Terms: conditions — Cicatrix; Acne Vulgaris

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Enlighten™ Laser and a MLA Attachment (Other): Enlighten™ Laser and a Micro-Lens Array Handpiece Attachment
  Interventions: Device: Enlighten™ Laser and a MLA Attachment

INTERVENTIONS:
Device: Enlighten™ Laser and a MLA Attachment — Subjects will receive treatments with the Cutera enlighten laser with the Micro-Lens Array handpiece attachment.

SUMMARY:
The purpose of this pivotal investigation is to evaluate the efficacy and safety of the Cutera enlighten multi-wavelength 532 nm and 1064 nm picosecond pulse duration laser and an investigational micro-lens array (MLA) handpiece attachment for improvement of moderate to severe acne scars.

DETAILED DESCRIPTION:
This is an open-label, prospective, multicenter, pivotal study in approximately 15 male or female subjects, age 18 to 65 years who desire laser treatment for the improvement of moderate to severe acne scars. Subjects will receive laser treatments with the Cutera enlighten laser with the Micro-Lens Array handpiece attachment. Subjects will return to the site after all study treatments have been delivered for a follow-up visit at 12 weeks following their final study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be able to read, understand and sign the Informed Consent Form.
2. Female or Male, 18 to 65 years of age (inclusive).
3. Fitzpatrick Skin Type I - VI.
4. Subject desires treatment for acne scars and wishes to undergo laser treatments for improvement.
5. Subject has bilateral moderate to severe signs of facial acne scarring.
6. Must be willing to have Cutera enlighten laser with the Micro-Lens Array handpiece attachment treatments and able to adhere to the treatments, follow-up visit schedule, and post-treatment care instructions.
7. Willing to have very limited sun exposure and use sunscreen on the treatment area every day for the duration of the study, including the follow-up period.
8. Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation (educational and/or marketing), publications, and any additional marketing purposes.
9. Agree to not undergo any other procedure(s) or treatment(s) for acne scars during the study and has no intention of having such procedures performed during the course of the study.
10. For female subjects: not pregnant or lactating and is either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study.,

Exclusion Criteria:

1. Participation in a clinical trial of another drug, or device administered to the treatment area, within 6 months prior to enrollment or during the study.
2. Any type of prior cosmetic treatment to the target area within 6 months of study participation, such as laser procedures, facial fillers, i.e. (Bellafill) and those used for general aesthetic correction, facial peel, lightening creams, or facial surgery.
3. Use of prescription topicals in the treatment area within one month prior to treatment or use of topical agents one week prior to treatment that may cause facial sensitivity.
4. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including but not limited to, open lacerations or abrasions, hidradenitis, rash, infection , or dermatitis of the treatment area prior to treatment (duration of resolution as per the Investigator's discretion).
5. Pregnant and/or breastfeeding, or planning to become pregnant.
6. Significant concurrent illness, such as diabetes mellitus, immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or using immunosuppressive medication.
7. Hypersensitivity to light exposure.
8. Any use of medication that is known to increase sensitivity to light according to the Investigator's discretion.
9. History of keloid scarring, hypertrophic scarring or abnormal wound healing or prone to bruising.
10. Has a history of squamous cell carcinoma or melanoma in the treatment area.
11. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity), including collagen vascular disease or vasculitic disorders.
12. A history or active skin condition that in the opinion of the Investigator may interfere/confound with the treatment.
13. History of connective tissue disease, such as systemic lupus erythematosus or scleroderma.
14. History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen.
15. History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation, or any that are considered not acceptable by the study investigator.
16. Has used oral isotretinoin (Accutane or therapeutic vitamin A supplements of ≥ 10,000 units per day) within 12 months of initial treatment or plans on using during the course of the study (note: skin must regain its normal degree of moisture prior to treatment, e.g. lack of noticeable skin flaking and peeling).
17. Excessively tanned or active sun tan in facial area to be treated, or unable/unlikely to refrain from tanning during the study.
18. Excessive facial hair in the area to be treated (beards, sideburns, and/or moustache,) that would interfere with diagnosis, assessment, and treatment.
19. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study, including excessive alcohol or drug abuses, or a condition that would compromise the subject's ability to comply with the study requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ronan, M.D., Principal Investigator — Cutera Research Center
Locations (1):
- Cutera Research Center, Brisbane, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enlighten™ Laser and a MLA Attachment
Started | 4
Completed | 2
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Enlighten™ Laser and a MLA Attachment
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Acne Scarring Improvement
Description: An improvement in Acne Scarring of at least one point on the Acne Scar Assessment Scale (ASAS):(1=clear scarring, 2=Very Mild scarring, 3=Mild scarring, 4=Moderate scarring or 5=Severe scarring) at the 12 weeks post final treatment
Time Frame: Baseline, and at 12 weeks post final treatment (up to 30 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enlighten™ Laser and a MLA Attachment
Number analyzed (Participants) | 2
score on a scale
  Baseline Acne Scar Assessment Scale Score | 4 (0)
  12 weeks post final treatment Acne Scar Assessment Scale Score | 4 (0)

ADVERSE EVENTS:
Time Frame: 12 weeks post-final treatment, up to 8 months
Arm/Group | Enlighten™ Laser and a MLA Attachment
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enlighten™ Laser and a MLA Attachment (N=4)
Erythema (Skin and subcutaneous tissue disorders) | 4
Edema (Skin and subcutaneous tissue disorders) | 2
Discomfort (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT03430921/Prot_001.pdf